CLINICAL TRIAL: NCT04177914
Title: Endoscopic Versus Shunt Treatment of Hydrocephalus in Infants
Brief Title: HCRN Endoscopic Versus Shunt Treatment of Hydrocephalus in Infants
Acronym: ESTHI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Alabama at Birmingham (Other); University of British Columbia (Other); University of Pittsburgh (Other); The Hospital for Sick Children (Other); Seattle Children's Hospital (Other); Vanderbilt University Medical Center (Other); Washington University School of Medicine (Other); Nationwide Children's Hospital (Other); Johns Hopkins University (Other); University of Calgary (Other); University of Colorado, Denver (Other); Children's Hospital Los Angeles (Other); National Institutes of Health (NIH) (NIH); Hydrocephalus Association (Other); Penn State University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Baylor College of Medicine (Other); University of Florida (Other); Orlando Health, Inc. (Other); Virginia Commonwealth University (Other); Trustees of Indiana University (Unknown)
Responsible Party: Principal Investigator, John Kestle, MD, Vice Chair of Clinical Research, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN 012; 1U01NS107486-01A1 (NIH)
Record Dates: First submitted 2019-10-27; First posted 2019-11-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; Infants; Ventriculoperitoneal Shunt; ETV+CPC; endoscopic third ventriculostomy; choroid plexus cauterization
MeSH Terms: conditions — Hydrocephalus | interventions — Ventriculostomy; Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETV+CPC (Active Comparator): Subjects randomized to this arm will undergo an ETV+CPC procedure for treatment of Hydrocephalus
  Interventions: Procedure: Endoscopic Third Ventriculostomy with Choroid Plexus Cauterization (ETV+CPC)
- Ventriculoperitoneal Shunt (Active Comparator): Subjects randomized to this arm will undergo a Ventriculoperitoneal Shunt procedure for treatment of Hydrocephalus
  Interventions: Device: Ventriculoperitoneal Shunt

INTERVENTIONS:
Procedure: Endoscopic Third Ventriculostomy with Choroid Plexus Cauterization (ETV+CPC) — Since the early 1990s, ETV has become the main alternative to shunting for hydrocephalus. This procedure involves placing an endoscopic camera into the ventricles of the brain and creating a hole in the floor of the third ventricle to act as an internal bypass for obstructed CSF. The cauterization of choroid plexus (CPC) involves the use of a device to burn or cauterize tissue from the choroid plexus. The choroid plexus of the brain exists in the lateral ventricles, the third ventricle, and the fourth ventricle. Its main role is the production of CSF. The success of ETV alone is poor in infants, but when combined with CPC, improved results have been observed and ETV+CPC has become a safe viable option for these children.
  Arms: ETV+CPC
Device: Ventriculoperitoneal Shunt — The most common treatment for hydrocephalus has been the insertion of a ventriculoperitoneal shunt, which has been in popular use for over 50 years. This consists of silastic tubing attached to a valve mechanism that runs subcutaneously from the head to the abdomen. It is one of the most common procedures performed by pediatric neurosurgeons.
  Arms: Ventriculoperitoneal Shunt

SUMMARY:
Hydrocephalus is a potentially debilitating neurological condition that primarily affects babies under a year of age and has traditionally been treated by inserting a shunt between the brain and the abdomen. A newer endoscopic procedure offers hope of shunt- free treatment that may reduce complications over a child's life, but it is not clear if the endoscopic procedure results in similar intellectual outcome as shunt. Therefore, the investigators propose a randomized trial to compare intellectual outcome and brain structural integrity between these two treatments, to help families make the best treatment decision for their baby.

DETAILED DESCRIPTION:
The ESTHI Trial is a multi-center randomized controlled trial (RCT) comparing endoscopic third ventriculostomy with choroid plexus cauterization (ETV+CPC) and shunt in infants with hydrocephalus. The study will leverage the infrastructure of the Hydrocephalus Clinical Research Network (HCRN), a committed group of 14 leading North American pediatric neurosurgical centers with a long track-record of successful collaborative clinical research and RCTs in hydrocephalus. Optimal cognitive outcome is the primary concern of families and will, therefore, be the primary outcome. Assessment of dMRI, a validated, non-invasive method of measuring white matter microstructural integrity and structural connectivity in the developing brain, will provide further insight into the developmental consequences of these two treatments. The results of the RCT will help families determine the optimal treatment of hydrocephalus for their child.

ELIGIBILITY:
Inclusion Criteria:

1. Corrected age <104 weeks and 0 days,

   AND
2. Child is ≥ 37 weeks post menstrual age,

   AND
3. Child must have symptomatic hydrocephalus, deﬁned as:

   Ventriculomegaly on MRI (frontal-occipital horn ratio (FOR) >0.45, which approximates "moderate ventriculomegaly"), and at least one of the following:
   * Head circumference >98th percentile for corrected age with either bulging fontanelle or splayed sutures
   * Upgaze paresis/palsy (sundowning)
   * CSF leak
   * Papilledema
   * Tense pseudomeningocele or tense ﬂuid along a track
   * Vomiting or irritability, with no other attributable cause
   * Bradycardias or apneas, with no other attributable cause
   * Intracranial pressure (ICP) monitoring showing persistent elevation of pressure with or without plateau waves

   AND
4. No prior history of shunt insertion or endoscopic third ventriculostomy (ETV) procedure (previous temporization devices and/or external ventricular drains permissible)

Exclusion Criteria:

1. Hydrocephalus due to intraventricular hemorrhage in a child born before 37 weeks gestational age; OR
2. Anatomy not suitable for ETV+CPC or anteriorly placed ventriculoperitoneal shunt deﬁned as:

   * Moderate to severe prepontine adhesions on steady state free precession (SSFP) or T2 weighted fast (turbo) spin echo (FSE/TSE) MRI, which includes the following sequences: FIESTA, FIESTA-C, TrueFISP, CISS, Balanced FFE (bFFE), CUBE, SPACE, VISTA, IsoFSE, and 3D MVOX
   * Closure of one or both foramina of Monro
   * Thick ﬂoor of third ventricle (≥ 3mm)
   * Narrow third ventricle (<5mm)
   * Presence of scalp, bone, or ventricular lesions that make placement of an anterior shunt impracticable; OR
3. Underlying condition with a high chance of mortality within 12 months; OR
4. Hydrocephalus with loculated CSF compartments; OR
5. Peritoneal cavity not suitable for distal shunt placement; OR
6. Active CSF infection; OR
7. Hydranencephaly; OR
8. Child requires an intraventricular procedure (e.g. endoscopic biopsy) in addition to the initial ﬁrst-time permanent procedure for the treatment of hydrocephalus.

Ages: 1 Day to 104 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Bayley Scale of Infant Development-IV (Bayley-IV) Cognitive Scale score | 12 months post randomized surgical intervention
  The primary objective is to determine, in infants <104 weeks corrected age, with hydrocephalus requiring treatment at tertiary care pediatric neurosurgery centers in North America, if treatment with ETV+CPC compared to shunt results in non-inferior cognitive outcome at 12 months from surgery, as measured by Bayley-IV Cognitive Scale score with a non-inferiority margin of 1.5. Scaled scores range from 1-19. Higher scores indicate better outcomes. Scores will also be obtained at 3 and 5 years of age.

SECONDARY OUTCOMES:
Bayley Scale of Infant Development-IV (Bayley-IV) Language Scaled Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Bayley-IV Language Scaled scores. Scaled scores range from 1-19. Higher scores indicate better outcomes.
Bayley Scale of Infant Development-IV (Bayley-IV) Motor Scaled Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Bayley-IV Motor Scaled scores. Scaled scores range from 1-19. Higher scores indicate better outcomes.

OTHER OUTCOMES:
Vineland-3 Communication Domain Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Vineland-3 Communication Domain scores. Domain scores range from 20-140. Higher scores indicate better outcomes.
Vineland-3 Daily Living Skills Domain Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Vineland-3 Daily Living Skills Domain scores. Domain scores range from 20-140. Higher scores indicate better outcomes.
Vineland-3 Socialization Domain Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Vineland-3 Socialization Domain scores. Domain scores range from 20-140. Higher scores indicate better outcomes.
Vineland-3 Motor Skills Domain Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Vineland-3 Motor Skills Domain scores. Domain scores range from 20-140. Higher scores indicate better outcomes.
Vineland-3 Adaptive Behavior Composite Score | 12 months post randomized surgical intervention
  To determine, in the same cohort of infants, if ETV+CPC compared to shunt results in non-inferior Vineland-3 Adaptive Behavior Composite (ABC) scores. ABC scores range from 20-140. Higher scores indicate better outcomes.
The occurrence of treatment failure. | Through study completion, a maximum of 7 years.
  Treatment failure is defined as obstruction, loculated compartments, overdrainage, CSF infection, or significant intraoperative complication. The rate of occurrence of each type, for the initial procedure, will be calculated. Failure can be captured at anytime during the course of the 7 year study. Occurrence between treatment arms will be compared.
Time to failure. | Through study completion, a maximum of 7 years
  Time to failure is the number of days in which the intervention is functionally successful. It is calculated from date of surgery to date of failure, as described in Outcome 9. Time to failure between treatment arms will be compared.
Total number of hospital admission days within 12 months after surgery | 12 months post randomized surgical intervention
  Number of days subject is admitted to the hospital during the first 12 months following the initial surgical intervention. All hospital admissions included, regardless of reason for admission. Number of hospital admission days between treatment arms will be compared.
Total number of repeat surgeries within 12 months after surgery | 12 months post randomized surgical intervention
  Number of shunt and ETV+CPC procedures during the first 12 months following the initial surgical intervention. Number of repeat surgeries between treatment arms will be compared.
Total number of brain imaging (CT, MRI, ultrasound) scans within 12 months after surgery | 12 months post randomized surgical intervention
  Number of CT, MRI, and ultrasound brain scans during the first 12 months following the initial surgical intervention. Total imaging between treatment arms will be compared.
All major peri-operative and post-operative complications | Through study completion, a maximum of 7 years
  Number of peri-operative and post-operative complications to include those related to CSF circulation, infection, hemorrhage, seizures, and new neurological deficits. Number of complications between treatment arms will be compared.
Brain and ventricle volume on MRI performed at 12 months after surgery | 12 months post randomized surgical intervention
  Brain and CSF volumes will be converted to Z-scores based on previously described age- and sex-adjusted distributions and used for comparison of brain volume and growth between ETV+CPC and shunt treatment groups.
dMRI corpus collosum (CC) and corticospinal tract (CST) fractional anisotropy (FA) at 12 months after surgery. | 12 months post randomized surgical intervention
  Develop dMRI maps, including fractional anisotropy (FA), mean diffusivity (MD), axial diffusivity (AD), and radial diffusivity (RD). Tract-based spatial statistics (TBSS) will be used for voxel-wise analyses of white matter tracts. Maps will be used to compare cerebral structural connectivity between the two treatment arms.
Cerebral spinal fluid myelin basic protein (MBP) levels measured at the time of ETV+CPC or shunt | 12 months post randomized surgical intervention
  Examine correlations of cerebral spinal fluid myelin basic protein (MBP) levels to post-operative Bayley-IV Cognitive Scale score.
Cerebral spinal fluid amyloid precursor protein (APP) levels measured at the time of ETV+CPC or shunt | 12 months post randomized surgical intervention
  Examine correlations of cerebral spinal fluid amyloid precursor protein (APP) to post-operative Bayley-IV Cognitive Scale score
Cerebral spinal fluid NCAM-1 levels measured at the time of ETV+CPC or shunt | 12 months post randomized surgical intervention
  Examine correlations of cerebral spinal fluid NCAM-1 levels to post-operative Bayley-IV Cognitive Scale score
Cerebral spinal fluid glial fibrillary acid protein (GFAP) levels measured at the time of ETV+CPC or shunt | 12 months post randomized surgical intervention
  Examine correlations of cerebral spinal fluid glial fibrillary acid protein (GFAP) to post-operative Bayley-IV Cognitive Scale score
Wechsler Preschool & Primary Scale of Intelligence (WPPSI) Scores | At 5 years of age
  To determine, in infants who reach 5 years of age before the end of the study, if ETV+CPC compared to shunt results in non-inferior WPPSI scaled scores. Scaled scores range from 1-19. Higher scores indicate better outcomes.
Health related quality of life (HRQoL) measurements | 12 months post randomized surgical intervention, and at 3 and 5 years of age
  To compare health-related quality of life (HRQoL), as measured by vi-sual analogue scales (VAS), Health Utilities Preschool (HuPS), and the Hydrocephalus Outcome Questionnaire (HOQ), between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: John Kestle, MD, Study Chair — University of Utah; Abhaya Kulkarni, MD, Principal Investigator — University of Toronto; David Limbrick, MD, Principal Investigator — Washington University School of Medicine; Richard Holubkov, PhD, Principal Investigator — University of Utah
Locations (21):
- United States (18):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Trustees of Indiana University, Indianapolis, Indiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - The Pennsylvania State University, University Park, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
After subject enrollment and 5 year follow up have been completed, we will prepare a final study database for analysis. A releasable database will be produced and completely de-identified in accordance with the definitions provided in the Health insurance Portability and Accountability Act (HIPAA). Namely, all identifiers specified in HIPAA will be recoded in a manner that will make it impossible to deduce or impute the specific identity of any patient. The database will not contain any institutional identifiers. We will also prepare a data dictionary that provides a concise definition of every data element included in the database. If specific data elements have idiosyncrasies that might affect interpretation or analysis, this will be discussed in the dictionary document.
  In accordance with policies determined by the investigators and funding sponsors, the releasable database will be provided to users in electronic form.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year of primary publication or within 18 months of the last study visit of the last subject, whichever occurs first.

DOCUMENTS (1):
  • Informed Consent Form (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04177914/ICF_000.pdf